CLINICAL TRIAL: NCT00779272
Title: Impact of Preoperative Chemotherapy on Complications and Regeneration After Resection of Colorectal Liver Metastases
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Breitenstein Stefan, Dr. med., Department Visceral and Transplantation Surgery, University Hospital of Zurich
Other Study IDs: StV 29-2008
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Colorectal Liver Metastases
Keywords: neoadjuvant chemotherapy; clinically postoperative outcome; liver regeneration after liver resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Without preoperative chemotherapy
- 2: With preoperative chemotherapy

SUMMARY:
The objective of this study is to evaluate for the first time not only the impact of neoadjuvant chemotherapy on clinical outcome, but also on liver regeneration after liver resection.

ELIGIBILITY:
Inclusion Criteria:

* Liver resection due to colorectal liver metastases between 2003 and 2007

Exclusion Criteria:

* Incomplete assessment of preoperative chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Records from 184 consecutive patients undergoing liver resection due to colorectal metastases between 2003 and July 2008 were reviewed from a prospective database
Sampling Method: Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Postoperative Complications and liver regeneration | 2003- July 2008

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Visceral and Transplantation Surgery of the University of Zurich, Zurich, Canton of Zurich, Switzerland